CLINICAL TRIAL: NCT00949351
Title: Safety of Add on Aliskiren to ACEI and ARB Treatment in Type 2 Diabetes With Nephropathy
Brief Title: Safety of Add on Aliskiren to Angiotensin Converting Enzyme Inhibitor (ACEI) and Angiotensin I Receptor Blocker (ARB) Treatment in Type 2 Diabetes With Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lerdsin General Hospital (Other)
Responsible Party: Division of Nephrology, Department of Medicine, Lerdsin General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lerdsin 36/52
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes With Nephropathy
Keywords: ACEI, ARB, DN, aliskiren, proteinuria
MeSH Terms: conditions — Proteinuria | interventions — aliskiren; Tacrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aliskiren (Placebo Comparator)
  Interventions: Drug: Aliskiren 300mg/d

INTERVENTIONS:
Drug: Aliskiren 300mg/d — Aliskiren 300mg/d v.s. placebo for 12wk
  Other Names: Rasilez (Thailand)

SUMMARY:
Activation of renin-angiotensin plays a crucial role diabetic nephropathy. Angiotensin converting enzyme inhibitor (ACEI) and Angiotensin I receptor blocker (ARB) has been shown renoprotection whether it was used alone or in combination. Aliskiren is a direct renin inhibitor (DRI) that has shown renal benefits and safety when combined with ARB. However, to date, the safety of add on aliskiren to the combination treatment of ACEI and ARB in diabetic nephropathy patients remains to elucidate.

ELIGIBILITY:
Inclusion Criteria:

* Type2 diabetes patients
* Age <30yrs-70yrs>
* Overt proteinuria (Urinary protein creatinine ratio > 200mg/g 2 times or more during past 6 Mo)
* Scr < 2.5 mg/dL
* HbA1C < 7.5
* Systolic blood pressure > 160 mmHg without antihypertensive drugs or > 140 with antihypertensive drug
* No history of previous cardiovascular event (Stroke, Myocardial infarction, unstable angina, hospitalization, surgical correction PVD or PVD with claudication)
* No hospitalization within 1 yr except for elective surgery

Exclusion Criteria:

* Physical examination found or suspected serious co-morbid (AF, carotid bruit, structural heart disease, cirrhosis and decompensate liver disease)
* Non adherence to protocol
* Intolerable to ACEI or ARB during run-in
* Abnormal liver function test at the run-in period
* Rapid declining renal function (SCr increase > 40%) during run-in
* Hyperkalemia (serum K > 5.5 mEq/L at randomization)
* Malignancy detected o
* SBP lower than 110 mmHg (at randomization)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-07 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Assess short-term safety of the combination of aliskiren 300 mg/valsartan 160 mg /enalapril 20 mg in patients with diabetic nephropathy | 12 wk after randomization

SECONDARY OUTCOMES:
Reduction of systolic blood pressure | 12 wk after randomization
Reduction of proteinuria | 12 wk after randomization
Change in GFR/mo | 12 wk after randomization
Change of Serum prorenin level compare to baseline | 12 wk after randomization
Change of Urinary TGFb1 compare to baseline | 12 wk after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Lerdsin General Hospital, Bangkok, Thailand